CLINICAL TRIAL: NCT05737589
Title: Integrated Circulating Tumor DNA and T Cell Repertoire Predict Radiotherapeutic Response and Outcome in Non-small Cell Lung Cancer Patients With Brain Metastasis
Brief Title: Circulating Tumor DNA and T Cell Repertoire Predict Radiotherapeutic Outcomes in NSCLC Patients With Brain Metastasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiaorong Dong (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Dong, Professor/Chief Physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: DTO-20230201
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Brain Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: This is an observational study, no interventions will be applied to patients in the observation group, and only blood and cerebrospinal fluid ctDNA and TCR data of patients with brain metastases from non-small cell lung cancer treated with radiotherapy will be recorded to predict patient prognosis. Peripheral blood and CSF samples were collected at baseline, 24 h (T0), and 28 days (T28) after completion of radiotherapy and underwent deep sequencing of ctDNA and TCR. The 6-month response rates of brain metastases and systemic lesions were evaluated based on Response Evaluation Criteria in Solid Tumors version 1.1 for further study.
  Interventions: Radiation: Whole-brain radiotherapy

INTERVENTIONS:
Radiation: Whole-brain radiotherapy — Radiotherapy is administered to the patient's brain lesions, and the subject's specific treatment plan is developed by two specialized physicians.
  Other Names: Stereotactic radiotherapy

SUMMARY:
Collection of ctDNA and TCR data to predict the efficacy and prognosis of brain radiotherapy in patients with brain metastases from non-small cell lung cancer (NSCLC) in a comprehensive manner

DETAILED DESCRIPTION:
The scarcity of biopsies or focal resections for brain metastases limits the discovery of biomarkers for diagnosing and prognosis of NSCLC patients with brain metastases. Circulating tumor DNA (ctDNA) is derived from the necrosis, apoptosis, and secretion of tumor cells and is widely distributed in various body fluids, including peripheral blood and cerebrospinal fluid (CSF). Genomic alterations in blood and CSF ctDNA are prognostic markers in NSCLC patients with brain metastases. Still, they have limited predictive power. T cell-mediated immune responses are essential to suppress carcinogenesis and metastasis in NSCLC. Targeted sequencing in the highly variable complementarity determining region 3 (CDR3) region of the T cell receptor (TCR) β-chain provides a powerful approach to quantifying the diversity of T cells. Radiotherapy causes antigen exposure through direct local destruction of cancer cells, which activates the local and systemic immune system. Radiotherapy can also cause intracellular DNA damage, and the ensuing mutations in DNA mismatch repair defects may increase neoantigen load, triggering an immune response. The TCR, closely related to immune system modifications, can also be altered by radiotherapy. However, no clinical studies have explored ctDNA and TCR to predict the efficacy and prognosis of brain radiotherapy in patients with NSCLC brain metastases. Therefore, we retrieved the visit data of 50 patients with advanced NSCLC brain metastases who received brain radiotherapy through the hospital electronic medical record system and recorded the ctDNA and TCR values of patients' blood and CSF at baseline (within 2 weeks before radiotherapy), T0 (within 24 hours after the completion of radiotherapy) and T28 (28 days after the completion of radiotherapy), disease progression recurrence and survival time by examining. The dynamic changes of ctDNA and TCR during brain radiotherapy were studied to comprehensively assess the ability of ctDNA and TCR to predict the efficacy and prognosis of brain radiotherapy in patients with NSCLC brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Patients must have histologically or cytologically confirmed NSCLC and imaging-confirmed primary non-small cell lung cancer with brain metastases
3. ECOG PS score of 0-2
4. At least 1 lesion meeting RECIST 1.1 target lesion (TL) criteria at baseline. Must have baseline assessment imaging of the tumor by CT or MRI scan within 28 days prior to treatment
5. No prior radiation therapy to the tumor, including but not limited to whole brain radiotherapy, prophylactic brain irradiation, stereotactic radiation therapy, etc.
6. Major organ function indicators meet the criteria for conventional radiation therapy Adequate organ and bone marrow function is defined as follows

   1. Hemoglobin ≥ 9.0 g/dL
   2. absolute neutrophil count ≥ 1.5 × 109 / L
   3. Platelet count ≥ 100 × 109 / L
   4. Serum bilirubin ≤ 1.5 × the upper limit of normal (ULN). The above criteria were not applied to patients diagnosed with Gilbert's syndrome, but these patients were allowed to be enrolled after consultation between the study physician and their primary care physician.
   5. Alanine aminotransferase ALT or aspartate aminotransferase AST ≤ 2.5 × ULN
   6. Creatinine clearance (CL) > 40 mL/min calculated or actually measured according to the Cockcroft-Gault method (based on actual body weight) Men. Creatinine CL = Body weight (kg) × (140 - age) (mL/min) 72 x serum creatinine (mg/dL) Females. Creatinine CL = Body weight (kg) × (140 - age) × 0.85 (mL/min) 72 × serum creatinine (mg/dL)
7. Female subjects of childbearing age must exclude pregnancy
8. Life expectancy >12 weeks
9. Body weight >30Kg

Exclusion Criteria:

1. History of allogeneic organ transplantation
2. Active or previously documented autoimmune or inflammatory disease (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis (except diverticular disease), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener's syndrome [granulomatous vasculitis, Graves' disease, rheumatoid arthritis, pituitary inflammation, uveitis, etc.])
3. History of active primary immunodeficiency
4. Other malignancies within the last 3 years.
5. Presence of uncontrolled co-morbidities including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmias, active interstitial lung disease, a severe chronic gastrointestinal disease with diarrhea or mental illness that limits compliance with study requirements, significantly increases the risk of AE or affects the patient's life/ social conditions
6. Active infection at the time of treatment, including tuberculosis (clinical assessment includes history, physical examination, imaging findings, and tuberculosis screening consistent with local clinical practice), hepatitis B (known hepatitis B surface antigen positive [HBsAg] result), hepatitis C virus (HCV) or human immunodeficiency virus (HIV 1/2 antibody positive). Patients with previous hepatitis B virus (HBV) infection or cured HBV infection (defined as the presence of positive hepatitis B core antibodies and negative HBsAg) may participate in this study. patients with positive HCV antibodies who are negative for HCV ribonucleic acid (RNA) by polymerase chain reaction only may participate in this study.
7. Stage IV NSCLC according to the 8th edition of the International Society for the Study of Lung Cancer Thoracic Oncology Staging Manual
8. Histological findings of NSCLC with mixed small cell component

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A group of non-small cell lung cancer patients with brain metastasis who have never received radiotherapy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-13 (Estimated); Primary Completion 2024-02-13 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | February 13, 2023-February 13, 2024
  OS is defined as the time elapsed between the initiation of radiotherapy and mortality from any cause.

SECONDARY OUTCOMES:
progression-free survival (PFS) | February 13, 2023-February 13, 2024
  PFS is defined as the time elapsed between the start of radiotherapy and the first sign of disease progression or death from any cause.
intracranial PFS (iPFS) | February 13, 2023-February 13, 2024
  The duration from the start of radiotherapy to the first intracranial lesion progression or death from any cause is referred to as iPFS.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Dong, Dr., Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
There is no data-sharing plan for other researchers.